CLINICAL TRIAL: NCT07184918
Title: Clinical Study Evaluating the Effect of Continuing or Discontinuing Angiotensin-Converting Enzyme Inhibitor on Renal Function in Patients Undergoing Coronary Angiography
Brief Title: Effect of Continuing vs. Discontinuing ACE Inhibitors on Renal Function After Coronary Angiography
Acronym: ACEI-RF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Magdy Ali Mohamed Radwan, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACEI-RF-2024
Record Dates: First submitted 2025-06-13; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Contrast-Induced Nephropathy; Coronary Angiography; Acute Kidney Injury
Keywords: CIN; Ramipril; Renal Function; Cardiac Catheterization; Nephrotoxicity; Renal Biomarkers
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Withholding Ramipril (Experimental): Discontinue Ramipril 48 hours prior to coronary angiograph.
  Interventions: Drug: Withholding Ramipril
- Arm 2: Continuing Ramipril (Active Comparator): Continue Ramipril throughout the peri-procedural period.
  Interventions: Drug: Continuing Ramipril

INTERVENTIONS:
Drug: Continuing Ramipril — Participants in this group will continue taking Ramipril at their usual dose before, during, and after the coronary angiography. The objective is to evaluate the renal effects of uninterrupted ACE inhibitor therapy during contrast exposure.
  Other Names: Tritace
  Arms: Arm 2: Continuing Ramipril
Drug: Withholding Ramipril — Participants in this group will stop taking Ramipril 48 hours before the angiography procedure and resume it 72 hours after. This intervention is used to evaluate whether temporarily withholding ACE inhibitors reduces the risk of contrast-induced nephropathy.
  Other Names: Tritace
  Arms: Arm 1: Withholding Ramipril

SUMMARY:
This clinical trial evaluates whether continuing or withholding ACE inhibitors (specifically Ramipril) before coronary angiography affects the risk of contrast-induced nephropathy (CIN). CIN is a known complication of iodinated contrast exposure, particularly in patients with chronic conditions such as hypertension or diabetes. The trial involves 44 adult patients randomized into two groups: one continuing Ramipril and the other withholding it 48 hours before and restarting 72 hours after the procedure. Renal biomarkers including serum creatinine, NGAL, and superoxide dismutase will be assessed to evaluate renal function.

DETAILED DESCRIPTION:
This randomized controlled study is designed to provide clinical evidence on whether withholding ACE inhibitors prior to contrast administration in coronary angiography affects kidney function. Participants are randomized into two arms: one arm will discontinue ACE inhibitors 48 hours prior and restart 72 hours post angiography, while the other will continue therapy without interruption. Primary endpoints include incidence of CIN as defined by a ≥0.5 mg/dL or ≥25% increase in serum creatinine within 72 hours. Secondary endpoints include NGAL, SOD, and potassium levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) scheduled for elective coronary angiography
* Currently on ACE inhibitor (Ramipril)
* Serum creatinine ≤1.5 mg/dL

Exclusion Criteria:

* STEMI within last 2 weeks
* NYHA Class IV heart failure
* CrCl <50 mL/min
* Serum potassium >5.0 mEq/L
* Recent contrast exposure
* Pregnancy or breastfeeding
* Cardiogenic shock or sepsis
* Severe uncontrolled hypertension

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Serum Creatinine at 72 Hours Post-Angiography | Baseline and 72 hours post-angiography
  CIN defined as ≥0.5 mg/dL or ≥25% rise in serum creatinine from baseline.

SECONDARY OUTCOMES:
Change in NGAL and SOD levels (pre vs post) | Baseline and 72 hours post-angiography
  Change in serum NGAL (Neutrophil Gelatinase-Associated Lipocalin) and SOD (Superoxide Dismutase) levels measured before and 72 hours after coronary angiography. These biomarkers are used to assess early tubular injury and oxidative stress respectively. Comparison will be made between intervention arms to determine whether ACE inhibitor withholding reduces renal cellular stress.
Incidence of Hyperkalemia After Coronary Angiography | Within 72 hours post-angiography
  Proportion of participants who develop hyperkalemia (defined as serum potassium >5.5 mmol/L) within 72 hours after coronary angiography. Comparison will be made between participants who continued ACE inhibitor therapy and those who withheld it to evaluate the impact of ACEI on electrolyte disturbance.
Incidence of Clinical Adverse Events Within 72 Hours | Within 72 hours post-angiography
  Occurrence of adverse clinical outcomes including dialysis requirement, myocardial infarction, stroke, or new-onset heart failure within 72 hours of coronary angiography. Events will be monitored and compared between the two intervention groups to evaluate safety related to ACE inhibitor continuation or withholding.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia R El-Afify, Assoc Prof, Study Chair — Tanta University
Locations (1):
- Faculty of Pharmacy Tanta university, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
The data collected in this study are part of a Master's thesis conducted at Tanta University. There is currently no plan to share individual participant data (IPD) due to institutional academic policies and ethical considerations.